CLINICAL TRIAL: NCT07292740
Title: Arthroscopic Glenoid Augmentation Using Upper Subscapularis Tendon In Recurrent Anterior Shoulder Dislocation
Brief Title: Arthroscopic Subscapularis Augmentation
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdellah Ammar Abdellah Morsy, principal investigator, Al-Azhar University
Other Study IDs: ASA
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The glenohumeral joint is the most commonly dislocated joint of the human body, The stability of GH joint relies on a complex network of static and dynamic structures.

Static stabilizers ::

DETAILED DESCRIPTION:
The glenohumeral joint is the most commonly dislocated joint of the human body, The stability of GH joint relies on a complex network of static and dynamic structures.

Static stabilizers ::

* include the congruency of the humeral head and glenoid, the glenoid labrum, glenohumeral ligaments surrounding the joint, and negative intra-articular pressure.

Dynamic stabilizers:

are primarily muscular and include the rotator cuff, which provides a compressive stabilizing effect, the tendon of the long head of the biceps, and muscles that stabilize the scapula ,The anterior labrum plays a key role in antero posterior stability as it deepens the glenoid cavity up to 50%.

anterior dislocation is the most common dislocation and is caused by the arm being positioned in an excessive amount of abduction and external rotation.

There are different methods of management

Can be achieved by several surgical techniques, according to whether the underlying etiology is a labral tear (Bankart) , humeral head lesion (Hill- Sachs) , or glenoid bone defect

Traumatic anterior shoulder instability without glenoid bone loss can be successfully treated with Bankart repair . On the other hand, bony procedures such as the Bristow and Latarjet procedures offer better outcomes in cases with concomitant glenoid bone loss greater than 21%-25% and engaging Hill-Sachs lesions

Controversy still exists regarding the ideal surgical treatment for AGI with limited (0%-13.5%) to subcritical (13.5%-25%) glenoid bone loss . Bony procedures are correlated with low recurrence, but high complication rates . On the contrary, clinical studies documented low complication rates [9], but higher recurrence rates or unsatisfactory outcomes for isolated or augmented Bankart repair in the context of subcritical glenoid bone loss

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients complaining of anterior glenoid instability , with 1 or more episodes of anterior shoulder dislocation.

  2. Associated limited (<13.5%) to subcritical (<25%) glenoid bone loss. 3. Positive anterior shoulder apprehension and pain refractory to conservative treatment.

  4. Age between (15 -49)years old

Exclusion Criteria:

* 1. Preexisting glenohumeral osteoarthritis, Infection 2. Multidirectional or voluntary shoulder instability. 3.. Acute proximal humerus fractures of the involved shoulder. 4.. refusable of patient

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: All patients were placed in the beach chair position after administration of general anesthesia or Regional anesthasia Diagnostic arthroscopy of the glenohumeral joint was The first step in accurate portal placement about the shoulder girdle is an identification of the subcutaneous anatomic landmarks; the scapular spine, acromial borders, AC joint, clavicle, and the coracoidprocess should b clearly identified. The posterior portal site can be localized as the (soft spot) in the triangular region between acromion, glenoid, andhumeral head; this point is variable but approximately 2 cm medial and 2 to 3 cm distal to the posterolateralcorner of the acromion
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Rowe score | 2nd and 6th months
  Assessment of the post operative and preoperative status of shoulder dislocation

REFERENCES:
- [Background] Dodson CC, Cordasco FA. Anterior glenohumeral joint dislocations. Orthop Clin North Am. 2008 Oct;39(4):507-18, vii. doi: 10.1016/j.ocl.2008.06.001. PMID 18803980
- [Background] Zhang M, Liu J, Jia Y, Zhang G, Zhou J, Wu D, Jiang J, Yun X. Risk factors for recurrence after Bankart repair: a systematic review and meta-analysis. J Orthop Surg Res. 2022 Feb 20;17(1):113. doi: 10.1186/s13018-022-03011-w. PMID 35184753